CLINICAL TRIAL: NCT05780164
Title: Improving Access and Recruitment to Clinical Trials for Lung Cancer Patients
Brief Title: Improving Access to Lung Cancer Clinical Trials
Acronym: Lung I-ACT
Status: Recruiting | Type: Observational
Sponsor: Oxford Brookes University (Other)
Collaborators: De Montfort University (Other)
Responsible Party: Principal Investigator, Dr Cathy Henshall, Reader in Nursing, Oxford Brookes University
Other Study IDs: IRAS Ref: 325757
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer; Patient Engagement; Research, Communication; Nurse-Patient Relations; Recruitment
Keywords: patient engagement; research, communication; clinical trials; nurse-patient relations; recruitment; lung cancer
MeSH Terms: conditions — Lung Neoplasms; Patient Participation; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Nurse participants will be provided with a research readiness tool to facilitate their discussions with lung cancer patients about clinical trial opportunities. The tool will be used by nurses over a six month period, alongside usual care.
  Interventions: Other: Research readiness tool
- Control: No intervention. Nurse participants will provide usual care to lung cancer patients.

INTERVENTIONS:
Other: Research readiness tool — Online/paper based tool containing information about lung cancer clinical trials
  Groups: Intervention

SUMMARY:
There are ~85,000 lung cancer patients (LCPs) in the UK; yet only around 8% were recruited into clinical trials in 2021/22. LCPs need opportunities to take part in clinical trials to access new treatments, increasing their quality of life, treatment choices and life expectancy.

Discussions with nurses can help patients make better treatment decisions, improving experiences of care. However, research has shown that lung cancer nurses (LCNs) often feel unable to discuss participation in trials with patients due to lack of knowledge, confidence, time and training.

This study aims to develop and test a research recruitment tool for LCNs, to support LCPs to enter clinical trials. Objectives include to:

* Explore reasons for low uptake of LCPs into clinical trials
* Develop a tool for LCNs to talk to patients about clinical trials
* Test whether the tool improves the number and quality of discussions nurses have with LCPs about clinical trials

The study has four phases:

Phase 1: A literature review will identify problems that make clinical trial uptake difficult for LCPs, carers and clinicians

Phase 2: Six group discussions with LCNs, patients and carers will explore issues that create potential barriers for patients taking part in clinical trials. The groups will take place online, last approximately one hour and be recorded.

Phase 3: Part 1&2 findings will help us develop a LCN research recruitment tool. The tool will contain information on how nurses obtain information about LC clinical trials, research teams, communication issues, practical issues and how to reach LCPs.

Phase 4: The research recruitment tool will be tested in four UK NHS hospitals. A survey will identify any changes in nurses' clinical trials awareness and confidence before and after using the tool. Interviews with LCNs, patients and carers will explore their views on the tool, clinical trials participation and experiences of care.

DETAILED DESCRIPTION:
Study design: This mixed methods study consists of the following phases:

Phase 1: systematic review exploring barriers and challenges to clinical trial uptake among LCPs, carers and clinicians

Phase 2: focus groups with LCPs, carers, LCNs, research nurses and multidisciplinary teams to explore challenges, barriers and facilitators to clinical trial uptake among LCPs

Phase 3: development of a research recruitment tool for LCNs to facilitate recruitment of LCPs into clinical trials Phase 4: pilot study to test the effectiveness and acceptability of the research recruitment tool across four NHS trusts (including interviews with LCPs, carers and LCNs).

Phase 1: A systematic review of the best scientific literature will identify challenges and barriers to clinical trial recruitment amongst LCPs, carers and clinicians. The research team have experience in conducting systematic reviews and share multi-disciplinary knowledge and expertise. A recent scoping exercise identified multiple papers examining recruitment to LC clinical trials; our review will be more extensive and rigorous in terms of databases searched, search terms, languages included, quality reviews of potential papers included and time period. PRISMA reporting guidelines will be followed.

Phase 2: Six qualitative focus groups with lung cancer patients, carers, lung cancer nurses and other members of the multidisciplinary team (MDT) will explore challenges and facilitators to LCPs' clinical trial entry. Focus group participants will be recruited through the participating sites lung cancer nursing teams.

Eligible clinician participants (nurses and other MDT staff) will be contacted through lead LCNs at participating sites (see phase 4), who will share invitation letters and participant information leaflets with their teams. These will explain the purpose of the study and provide details of what is involved. The letter will include the contact details of the research team and nurse participants will be asked to contact them if they are interested in taking part. A member of the research team will then offer to speak to the participants if they have any further questions about the study. If they are still happy to proceed the researcher will organise a time, date and place with participants to proceed with the focus group. Participants will also be recruited through LCNUK and the National Institute for Health Research (NIHR) Local Clinical Research Networks, who will provide access to an online link where potential participants can access information about the study (PIS and invitation letter) and can sign up via an online consent platform. Once consented the research team will contact them about the study and confirm they are happy to take part.

Patients and carers will be eligible to take part if they meet the following eligibility criteria:

Patients and carers will be recruited through the NCRI consumer forum and other cancer patient/carer networks, including RCLCF and Mesothelioma UK, who will provide access to an online link where potential participants can access information about the study (PIS and invitation letter) and can sign up via an online consent platform. Once consented the research team will contact them about the study and confirm they are happy to take part. LCNs at participating NHS sites will share invitation letters and information leaflets with LCPs, inviting them to take part. These will explain the purpose of the study and provide details of what is involved. The letter will include the contact details of the research team and nurse participants will be asked to contact them if they are interested in taking part. A member of the research team will then offer to speak to the participants if they have any further questions about the study. If they are still happy to proceed the researcher will organise a time, date and place with participants to proceed with the focus group. The study will also be promoted via social media channels such as Twitter. We intend to recruit ~48 participants to focus groups (eight per group); three focus groups will be with LCNs, research nurses and multidisciplinary team members from district general hospitals (DGHs) and tertiary centres, and two with LCPs and carers. A final group will include clinicians from the Christie and Royal Marsden cancer centres, where recruitment to trials is higher than in DGHs and tertiary centres, to identify transferable elements of best practice. Team members are affiliated with participating NHS sites and will utilise local contacts to facilitate recruitment. A topic guide will explore issues around LC trials awareness, knowledge of referral processes, confidence discussing trials, communication networks, time issues and factors influencing trial entry. Focus groups will be held virtually via Microsoft Teams. Participants will provide online consent and demographic information. Focus groups facilitated by two researchers, will last one hour, and will be recorded and transcribed. Data will be thematically analysed using the Framework Method, to enable comparisons across groups to be identified and themes generated [20].

Phase 3: Phase 1&2 findings will inform development of the LCN research recruitment tool. The tool, available in paper and online formats, will include information on finding out about LC clinical trials, the role of research teams, embedding research into multidisciplinary team meetings and health needs assessments, communication pathways, signposting LCPs, practical considerations and reaching underrepresented groups. Tool development will be guided by the Trial Steering Group (TSG), with representation from LC patient and public involvement (PPI) members, LCNs, multidisciplinary research and clinical teams. The tool will be tested for face and content validity by ~10 LCNs who participated in Phase 2, and ~4 PPI representatives. Relevant feedback will be used to make modifications to the tool.

Phase 4 pilot: Participants in the pilot study will pilot the research recruitment tool for proof of concept across four UK NHS sites, including tertiary centres and DGHs: Oxford, Derby&Burton, Lanarkshire, Nottinghamshire. An additional two NHS sites, Surrey and Birmingham, will act as controls.

Each site's LCNs (n=36) will be invited to participate through their senior nurse manager who will provide eligible nurses with an online invitation letter and participant information sheet (PIS). This will explain the purpose of the study and provide details of what is involved. The letter will include the contact details of the research team and nurse participants will be asked to contact them if they are interested in taking part. A member of the research team will then offer to speak to the participants if they have any further questions about the study. If they are still happy to proceed the researcher will organise a time, date and place with participants to proceed with the pilot phase of the study. Nurse participants will then have a briefing session, where the pilot study purpose will be explained. LCNs at the pilot sites (n=24) will be provided with a training session on using the tool, before implementing it in their teams for six months. Survey data will be collected from each LCN (n=36) at baseline, three and six months and LCN's will reconsent electronically, via the Qualtrics survey platform, prior to completing each online survey. The survey will collect information on the following: 1) Items from the validated General Perceived Self-Efficacy Scale will measure LCNs' self-efficacy (primary outcome measure) in relation to their research roles 2) The number of LCPs each LCN has approached to discuss clinical trial opportunities will be recorded 3) Likert style survey data on LCNs' knowledge, confidence and awareness of clinical trials will be collected. These questions will be developed from phase 1&2 findings and tested for reliability and validity by TSG members. The repeated tests measure ANOVA will compare survey responses between baseline, three and six months. Between groups ANOVA will compare differences in scores between pilot and control sites. No formal sample size calculation is required as this is a pilot study; however, all LCNs across the six sites will be invited to take part (n~36). Towards the end of the pilot, eight LCNs who have been taken part in the pilot will be invited, via an invitation letter and participant information sheet provided by the research team, to attend a 30-minute interview to explore the tool's acceptability, in terms of ease of use and impact on recruitment. We intend to invite between 1-2 nurses from each site to take part in the interview and they will be convenience sampled. Eight patients/carers who have joined clinical trials at the pilot sites will also be interviewed.

Patients and carers will be recruited through the LCNs and RCLCF and Mesothelioma UK networks, who will facilitate contact with local LCP support groups. LCP and carers clinical trial experience and its impact on quality of life, care satisfaction, self-efficacy and symptom control will be explored. This will provide valuable information on the tool's impact on LCP experience.

Ethics: NHS HRA ethics will be obtained, as well as local R&D approvals from each of the participating NHS Trust sites prior to recruitment commencing at these sites. Participants will be given detailed information sheets covering all relevant aspects of their involvement in the project, including confidentiality and GDPR. All participants will be asked to sign a consent form. Project team members and facilitators all understand the principles of safeguarding. Specifically, they will: understand they have a duty of care for and a responsibility to protect the health, wellbeing and human rights of participants; recognise participants may be at increased risk of distress due to the nature of the study; understand how to offer practical and emotional support; know how to signpost to any relevant support services.

Reporting and Future Research Ideas and recommendations generated through a discussion of the findings will be used to inform best practice and to implement clinical standards across the NHS. They will be reported in peer-reviewed publications and presented at conferences. A summary report of findings will be published on the University's website, as well as on the Roy Castle Lung Cancer Foundation website to ensure availability to patients and the public. In addition, findings will be promoted and disseminated through our partners Lung Cancer Nursing UK, Mesothelioma UK, Scottish Lung Cancer Nursing Forum, National Cancer Research Institute and British Thoracic Oncology Group, as well as via social media channels.

Following completion of the project, the project team will review the potential for the research readiness tool that has been developed to be implemented and evaluated across a larger number of NHS sites, with recommendations for the tool's use being generated, to inform policy and practice in this area.

Timelines: The timeline for the project is 24 months, including the time taken to obtain relevant permissions and approvals prior to the commencement of the interview study. It is anticipated that survey, focus group and interview recruitment, data collection and analysis will take be carried out from Oct 2023 to March 2025, and the reporting and dissemination will take place from April to June 2025. Four six monthly steering group meetings are planned throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurse with Nursing and Midwifery Council
* Actively involved in the clinical care pathways of lung cancer patients
* Working at one of the six participating NHS trusts
* Age between 18-65 years of age

Exclusion Criteria:

* Not actively involved in frontline clinical care
* Not involved in caring for lung cancer patients for at least 30% of their role
* Employed as a lung cancer research delivery nurse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients, carers and healthcare professionals
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived self-efficacy of nurses ability to discuss clinical trials with lung cancer patients | Data will be collected from each LCN (n=36) at baseline, three and six months.
  Items from the validated General Perceived Self-Efficacy Scale will measure lung cancer nurses' self-efficacy in relation to their research.
Perceived self-efficacy of nurses ability to discuss clinical trials with lung cancer patients | Data will be collected from each LCN (n=36) at three months.
  Items from the validated General Perceived Self-Efficacy Scale will measure lung cancer nurses' self-efficacy in relation to their research.
Perceived self-efficacy of nurses ability to discuss clinical trials with lung cancer patients | Data will be collected from each LCN (n=36) at six months.
  Items from the validated General Perceived Self-Efficacy Scale will measure lung cancer nurses' self-efficacy in relation to their research.

SECONDARY OUTCOMES:
number of Lung cancer patients each nurse has approached to discuss clinical trial opportunities | Data will be collected from each Lung Cancer Nurse (n=36) at baseline.
  Data willl be collected on number of times nurses have discussed trials opportuniites with patients
number of Lung cancer patients each nurse has approached to discuss clinical trial opportunities | Data will be collected from each Lung Cancer Nurse (n=36) at three months.
  Data willl be collected on number of times nurses have discussed trials opportuniites with patients
number of Lung cancer patients each nurse has approached to discuss clinical trial opportunities | Data will be collected from each Lung Cancer Nurse (n=36) at six months
  Data willl be collected on number of times nurses have discussed trials opportuniites with patients
Nurses' knowledge, confidence and awareness of clinical trials | Data will be collected from each LCN (n=36) at baseline.
  Likert style survey data
Nurses' knowledge, confidence and awareness of clinical trials | Data will be collected from each LCN (n=36) at three months.
  Likert style survey data
Nurses' knowledge, confidence and awareness of clinical trials | Data will be collected from each LCN (n=36) at six months.
  Likert style survey data

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Henshall, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Faculty of Health and Life Sciences, Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared woith researchers outside of the study team. Hwever, deidentified data will be shared through publications and reports and other dissemination activities.